CLINICAL TRIAL: NCT03493490
Title: Neodolpasse® Infusion Solution Versus Diclofenac 75 mg Infusion in the Treatment of Postoperative Pain After Elective Knee Surgery - an Exploratory Placebo-controlled Clinical Study to Investigate the Analgesic Properties of the Combination of Diclofenac and Orphenadrine Versus Diclofenac Alone.
Brief Title: Neodolpasse® Infusion Solution Versus Diclofenac 75 mg Infusion in the Treatment of Postoperative Pain After Elective Knee Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Oliver Kimberger, Deputy Head of Department of Anesthesiology, General Intensive Care and Pain Medicine, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NDOL-001-2016
Record Dates: First submitted 2018-03-16; First posted 2018-04-10 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative; Analgesic Adverse Reaction; Cruciate Ligament Rupture
Keywords: Double-Blind Method; placebo-controlled; parallel-group; single-centre; exploratory clinical study
MeSH Terms: conditions — Pain, Postoperative | interventions — Neodolpasse; Diclofenac

STUDY DESIGN:
Intervention Model Description: Randomization of the study patient takes place pre-surgery. Successfully randomized patients will receive two infusions over 30 minutes after fixation of the graft replacement and with a time interval of 8 hours each during the first 24 hours postoperatively. All patients will be provided with a PCA device as postoperative rescue medication. Consequently the possibility of an inadequate postoperative pain treatment in the study patients is very low, also in the placebo group.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neodolpasse (Experimental): In the Neodolpasse® arm patients receive two infusions over 30 minutes after fixation of the graft replacement and with a time interval of 8 hours each during the first 24 hours.
  Neodolpasse® Infusion Solution combines 75 mg (250 mL) of the NSAID diclofenac with 30 mg of the muscle-relaxant orphenadrine.
  Interventions: Drug: Neodolpasse
- Diclofenac (Active Comparator): In the Diclofenac arm patients receive two infusions over 30 minutes after fixation of the graft replacement and with a time interval of 8 hours each during the first 24 hours.
  The Infusion solution contains 75 mg (250 mL) of the NSAID diclofenac.
  Interventions: Drug: Diclofenac
- Placebo (Placebo Comparator): In the Placebo arm patients receive two physiologic saline infusion (250 mL) over 30 minutes after fixation of the graft replacement and with a time interval of 8 hours each during the first 24 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neodolpasse — Patients will receive two infusions containing 75 mg diclofenac and 30 mg orphenadrine citrate 30 minutes after fixation of the graft replacement and with a time interval of 8 hours.
  Arms: Neodolpasse
Drug: Diclofenac — Patients will receive two infusions containing 75 mg diclofenac 30 minutes after fixation of the graft replacement and with a time interval of 8 hours.
  Arms: Diclofenac
Drug: Placebo — Patients will receive two physiologic saline infusions 30 minutes after fixation of the graft replacement and with a time interval of 8 hours.
  Arms: Placebo

SUMMARY:
The clinical study is planned as a double-blind, randomised, placebo-controlled, parallel-group, single-centre exploratory clinical study with the aim to investigate the analgesic efficacy of the Neodolpasse® Infusion Solution in comparison to a 75 mg diclofenac only infusion. Included will be Patients receiving elective cruciate ligament surgery. The effectiveness will be measured by the use of additional analgesic medication via PCA during the first 24 hours postoperatively as well as by using a Visual Analogue Scale (VAS). Furthermore the local and systemic tolerability and safety of the clinical study medications (i.e. Neodolpasse® Infusion Solution and 75 mg diclofenac only infusion) will be assessed.

DETAILED DESCRIPTION:
The clinical study is planned as a double-blind, randomised, treatment-controlled, parallel-group, single-centre exploratory clinical study with the aim to investigate the analgesic efficacy of the Neodolpasse® Infusion Solution in comparison to a 75 mg diclofenac only infusion.

Patients who meet the inclusion and exclusion criteria will be enrolled to the clinical study and receive an enrolment number. The enrolment number will be a 4-digit number where the leftmost position will be zero ("0"). Enrolled patients will receive enrolment numbers starting at 0001, 0002, and so forth.

Only patients who were successfully randomized after surgery will continue the study protocol. All other patients will be regarded as screening failures. Successfully randomized patients will receive two infusions over 60 - 90 minutes with a time interval of 8 hours each during the first 24 hours postoperatively. All patients will be provided with a PCA device and will be allowed on demand analgetics as postoperative rescue medication. Consequently the possibility of an inadequate postoperative pain treatment in the study patients is very low.

Anaesthesia will be induced with propofol (1.0-2.5 mg/kg), remifentanil (1 mcg/kg over minimum of 30s) and rocuronium (0.6mg/kg) and subsequently maintained with remifentail (0.25 - 1 mcg/kg/min), and sevoflurane. During skin suture, 7.5 mg piritramid will be administered. No nitrous oxide will be administered.

No other narcotics, analgesics, or sedatives than those described herein will be allowed. In case the surgical procedure mandates the use of additional and/or other narcotics, analgesics, or sedatives it shall be up to the investigator to decide on further treatment. However, in such case the patient will not be randomized and will be regarded as screening failure.

Randomization of the study patient takes place post-surgery as soon as the patient is able to cooperate adequatey. Ability to cooperate is defined as successful VAS assessment. At this time point the patient will be randomized and assigned her/his final randomisation number. The final randomisation number will be a 4-digit number where the leftmost position indicating the type of knee surgery performed. Patient undergoing surgery for cruciate ligament repair will receive randomisation numbers starting at 1001, 1002, and so forth. Patients undergoing knee replacement surgery will receive randomisation numbers starting at 2001, 2002, and so forth.

The first infusion of the investigational medicinal product will be started immediately after randomization. PCA will be established as soon as possible after the start of the first infusion of the investigational medicinal product but not later than 30 min after the start of the first infusion of the investigational medicinal product. A one-way PCA device (Vygon PCA-System) will be used. The PCA system is independent from any power supply and therefore both safe and reliable. The PCA system contains 20 mg Hydal® (hydromorphone) in 50 mL solvent. The PCA system parameters are fixed to a single bolus volume of 0.5 mL thus delivering 0.2 mg hydromorphone per bolus which equates to 2.0 mg piritramide or 1.5 mg morphine. Lock-out period of the PCA system used is fixed to 5 min.

All bolus injections will be recorded and added to the cumulative analgesic doses delivered by PCA.

ELIGIBILITY:
Inclusion Criteria:

* Elective cruciate ligament surgery
* Confirmed patient suitability for planned surgery
* Legally valid signed written informed consent provided
* Female patients are confirmed non-pregnant (negative pregnancy test) or not breast feeding
* Adequate renal function defined by a creatinine value lower than 1.80 mg/dL for male and ower than 1.50 mg/dL for female patients
* No known intolerabilities or hypersensitivities to any part of the IMP / control medication
* No reoperation/revision within 6 months after the initial surgery
* Absence of history of abuse of analgesics or other drug
* No analgesics within 48 hours prior to surgery (surgery-related medication excluded)
* No current / recent (within 4 weeks prior to enrolment) experimental treatment
* No current / recent (within 4 weeks prior to enrolment) participation in another clinical study
* No foreseeable difficulties with regard to protocol compliance
* No known hypersensibility against the active ingredients diclofenac, orphenadrine, remifentanil, propofol, rocuronium, and hydromorphone
* No known hypersensibility against the other ingredients of the investigational medicinal product
* Absence of congestive heart failure classes 2 or higher according to the NYHA classification
* Absence of ischemic heart disease
* Absence of peripheral arterial occlusive disease
* Absence of cerebro-vascular disease
* Absence of significant risk factors for cardiovascular events (e.g., hypertension, hyperlipidaemia, type-2 diabetes, moderate smoking defined as consumation of 11 cigarettes or more per day)

exclusion criteria

* Major complications during surgery possibly leading to problems in the handling of the PCA or subsequently with the experimental treatment
* Intolerable adverse events or any serious adverse event
* Severe violation of the clinical study protocol
* Withdrawal of patient informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
PCA-use: Total dose of PCA alangetics required over the first 24 hours post-surgery. Measured in mg | within 24 hours
  amount of pca analgetic administered

SECONDARY OUTCOMES:
VAS-Scale: Pain relief will be tracked during the infusion periods and until 48 hours after the surgical intervention by using a Visual Analogue Scale (VAS). | after 24 hours
  visual analogue scales (VAS) pain measured The pain VAS is a unidimensional measure of pain intensity, used to record patients' pain pain severity. The VAS used is a straight horizontal line of fixed length 100 mm and pople scored their Pain 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Kimberger, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jin F, Chung F. Multimodal analgesia for postoperative pain control. J Clin Anesth. 2001 Nov;13(7):524-39. doi: 10.1016/s0952-8180(01)00320-8. PMID 11704453
- [Background] Kehlet H. Synergism between analgesics. Ann Med. 1995 Apr;27(2):259-62. doi: 10.3109/07853899509031968. PMID 7632423
- [Background] Kornhuber J, Parsons CG, Hartmann S, Retz W, Kamolz S, Thome J, Riederer P. Orphenadrine is an uncompetitive N-methyl-D-aspartate (NMDA) receptor antagonist: binding and patch clamp studies. J Neural Transm Gen Sect. 1995;102(3):237-46. doi: 10.1007/BF01281158. PMID 8788072
- [Background] Hunskaar S, Berge OG, Hole K. Orphenadrine citrate increases and prolongs the antinociceptive effects of paracetamol in mice. Acta Pharmacol Toxicol (Copenh). 1986 Jul;59(1):53-9. doi: 10.1111/j.1600-0773.1986.tb00134.x. PMID 3766151
- [Background] Luetz A, Heymann A, Radtke FM, Chenitir C, Neuhaus U, Nachtigall I, von Dossow V, Marz S, Eggers V, Heinz A, Wernecke KD, Spies CD. Different assessment tools for intensive care unit delirium: which score to use? Crit Care Med. 2010 Feb;38(2):409-18. doi: 10.1097/CCM.0b013e3181cabb42. PMID 20029345